CLINICAL TRIAL: NCT01798056
Title: An Observer-blind Study to Evaluate Immunogenicity and Safety of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A in Adults 18 Years of Age or Older With Solid Tumours Receiving Chemotherapy
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Herpes Zoster (HZ/su) Vaccine in Adults With Solid Tumours Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 116427; 2012-002966-11 (EudraCT Number)
Record Dates: First submitted 2013-02-14; First posted 2013-02-25 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Herpes Zoster; Herpes Zoster Vaccine
Keywords: ≥18 years of age; Chemotherapy; Solid tumours; Immunogenicity; Herpes Zoster; Safety; Shingles
MeSH Terms: conditions — Herpes Zoster | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- GSK1437173A Group (Experimental): Subjects received the first dose of GSK 1437173A at least 10 days (up to 1 month) before start of chemotherapy cycle or at the first day (allowing a window of +/- 1 day) of the first (or second) chemotherapy cycle. The second dose of GSK 1437173A vaccine was administered between 1 and 2 months after the first vaccination and at the first day (allowing a window of +/- 1 day) of a subsequent cycle of chemotherapy. The study products were administered intramuscularly into a deltoid muscle. The choice of and use of chemotherapy, or any other medication related to the patients' current conditions, were based on the local standard of care for the patients.
  Interventions: Biological: GSK 1437173A
- Placebo Group (Placebo Comparator): Subjects received the first dose of placebo at least 10 days (up to 1 month) before start of chemotherapy cycle or at the first day (allowing a window of +/- 1 day) of the first (or second) chemotherapy cycle. The second dose of placebo was administered between 1 and 2 months after the first vaccination and at the first day (allowing a window of +/- 1 day) of a subsequent cycle of chemotherapy. The study products were administered intramuscularly into a deltoid muscle. The choice of and use of chemotherapy, or any other medication related to the patients' current conditions, were based on the local standard of care for the patients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: GSK 1437173A — 2 doses administered by intramuscular (IM) injection into the deltoid muscle of the non-dominant arm.
  Other Names: HZ/su; GSK Biologicals Herpes Zoster subunit (HZ/su) vaccine
  Arms: GSK1437173A Group
Drug: Placebo — 2 doses administered by IM injection into the deltoid muscle of the non-dominant arm.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of GSK Biologicals' HZ/su vaccine in adults with solid tumours undergoing chemotherapy.

DETAILED DESCRIPTION:
The study will be randomised into two groups based on the vaccination schedule in relation to the start of a chemotherapy cycle:

* The OnChemo group receives their first HZ/su vaccination at the start of a chemotherapy cycle,
* The PreChemo group receives their first HZ/su vaccination at least 10 days before the start of a chemotherapy cycle.

The protocol summary has been updated following Protocol Amendment 2, August 2014, leading to the increase of the enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* A male or female aged 18 years or older (and has reached the age of legal consent) at the time of study entry (i.e., when informed consent is signed).
* Subject who has been diagnosed with one or more solid tumours (defined as a solid malignancy, i.e., not a blood element malignancy).
* Subject who is receiving or will receive a cytotoxic or immunosuppressive chemotherapy (such that the study vaccine can be administered at the latest at the start of the second cycle of chemotherapy).
* Life expectancy of greater than one year.
* Female subjects of non-childbearing potential may be enrolled in the study:

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause;
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Subjects receiving only newer, more targeted therapies if not taken together with a classical chemotherapy.
* Chronic administration and/or planned administration of systemic glucocorticoids within one month prior to the first vaccine dose and up to Visit 3 (Month 2). Inhaled, intra-articularly injected, and topical steroids are allowed.
* Previous vaccination against HZ or varicella within 12 months preceding the first dose of study vaccine/ placebo.
* Planned administration during the study of a HZ vaccine (including an investigational or non-registered vaccine) other than the study vaccine.
* Previous chemotherapy course less than one month before first study vaccination.
* Occurrence of a varicella or HZ episode by clinical history within the 12 months preceding the first dose of study vaccine/ placebo.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine or study material and equipment.
* Administration or planned administration of a live vaccine in the period starting 30 days before the first dose of study vaccine and ending 30 days after the last dose of study vaccine, or, administration or planned administration of a non-replicating vaccine within 8 days prior to or within 14 days after either dose of study vaccine.
* HIV infection by clinical history.
* Acute disease and/or fever at the time of vaccination. Acute disease is defined as the presence of a moderate or severe illness with or without fever, but excludes the underlying malignancy, as well as the expected symptoms/signs associated with that disease or its treatment:

  * Fever is defined as temperature ≥ 37.5°C /99.5°F on oral, axillary or tympanic setting, or ≥ 38.0°C /100.4°F on rectal setting. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever, may receive the first dose of study vaccine/ placebo at the discretion of the investigator.
* Any condition which, in the judgment of the investigator would make intramuscular injection unsafe.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions (if of childbearing potential) before Month 3 (i.e., 2 months after the last dose of study vaccine/ placebo).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2015-06-18 (Actual); Study Completion 2016-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- Canada (3):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Prague, Czechia
- France (4):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Férolles-Attilly
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Nîmes
- GSK Investigational Site, Seoul, South Korea
- Spain (7):
  - GSK Investigational Site, Badajoz
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Móstoles
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, San Sebastián de los Reyes
- United Kingdom (6):
  - GSK Investigational Site, Cheltenham, Gloucestershire
  - GSK Investigational Site, Woolwich, London
  - GSK Investigational Site, Swindon, Wiltshire
  - GSK Investigational Site, Exeter
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, York

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=114720

REFERENCES:
- [Background] Vink P, Delgado Mingorance I, Maximiano Alonso C, Rubio-Viqueira B, Jung KH, Rodriguez Moreno JF, Grande E, Marrupe Gonzalez D, Lowndes S, Puente J, Kristeleit H, Farrugia D, McNeil SA, Campora L, Di Paolo E, El Idrissi M, Godeaux O, Lopez-Fauqued M, Salaun B, Heineman TC, Oostvogels L; Zoster-028 Study Group. Immunogenicity and safety of the adjuvanted recombinant zoster vaccine in patients with solid tumors, vaccinated before or during chemotherapy: A randomized trial. Cancer. 2019 Apr 15;125(8):1301-1312. doi: 10.1002/cncr.31909. Epub 2019 Feb 1. PMID 30707761
- [Derived] Hirsch C, Zorger AM, Baumann M, Park YS, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with solid tumours. Cochrane Database Syst Rev. 2025 Apr 16;4(4):CD015551. doi: 10.1002/14651858.CD015551.pub2. PMID 40237463
- See also: Full CSR posting on gsk. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=116427&attachmentIdentifier=bf67d7ed-58e4-4f70-8a4d-0a418b627542&fileName=gsk-116427-clinical-study-report-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 237 subjects initially enrolled in the study, only 232 subject were included in the Total Vaccinated Cohort.
Period: Overall Study
Arm/Group | GSK1437173A Group | Placebo Group
Started | 117 | 115
Completed | 90 | 90
Not Completed | 27 | 25
Not completed — Serious Adverse Event | 13 | 12
Not completed — Withdrawal by Subject | 12 | 9
Not completed — Migrated/moved from study area | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1437173A Group | Placebo Group | Total
Number analyzed (Participants) | 117 | 115 | 232
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (10.8) | 58.5 (11.7) | 57.79 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 69 | 139
  Male | 47 | 46 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage/African American | 2 | 2 | 4
  Geographic ancestry: American Indian or Alaskan Native | 2 | 0 | 2
  Geographic ancestry: Asian - East Asian Heritage | 11 | 14 | 25
  Geographic ancestry: Asian - South East Asian Heritage | 0 | 2 | 2
  Geographic ancestry: White - Arabic/North African Heritage | 1 | 0 | 1
  Geographic ancestry: White - Caucasian/European Heritage | 92 | 88 | 180
  Geographic ancestry: Mixed Origin | 0 | 1 | 1
  Geographic ancestry: Missing | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Geometric Means for Anti-glycoprotein E (gE) Antibodies in PreChemo Groups
Description: Adjusted geometric means (GMC) of GSK1437173A over placebo for anti-glycoprotein E (gE) antibody enzyme-linked immunosorbent assay (ELISA) concentrations in PreChemo Groups only.
Time Frame: At Month 2
Population: The analysis was performed on the PreChemo groups from the According-to-Protocol (ATP) cohort for Humoral immunogenicity which included all evaluable subjects up to 30 days post last vaccination and who had met all eligibility criteria and complied with the procedures and intervals defined in the protocol for active phase of the study.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Groups:
- GSK1437173A-PreChemo: Subjects receiving the adjuvanted GSK1437173A vaccine, with the first vaccination at least 10 days (up to 1 month) before the start of a chemotherapy cycle. The choice of and use of chemotherapy, or any other medication related to the patients' current conditions, were based on the local standard of care for the patients.
- Placeb-PreChemo: Subjects receiving saline placebo, with the first vaccination at least 10 days (up to 1 month) before the start of a chemotherapy cycle. The choice of and use of chemotherapy, or any other medication related to the patients' current conditions, were based on the local standard of care for the patients.
Arm/Group | GSK1437173A-PreChemo | Placeb-PreChemo
Number analyzed (Participants) | 65 | 76
EL.U/mL | 24501.57 [19051.99 to 31509.94] | 1056.77 [990.37 to 1127.62]
Statistical Analysis 1: Comparison: GSK1437173A-PreChemo vs Placeb-PreChemo; The analysis evaluated the anti-gE humoral immune responses at Month 2, following a two-dose administration of the GSK1437173A vaccine, as compared to placebo in subjects with solid tumours receiving chemotherapy (PreChemo Groups only); Test type: Non-Inferiority — Criteria used: The lower limit (LL) of the 95% confidence interval (CI) of the Geometric Mean (GM) ratio (GSK1437173A PreChemo group over Placebo PreChemo group) in anti-gE ELISA antibody concentrations is greater than 3; Difference of means between vaccines and placebo were calculated together with 2-sided confidence intervals and back-transformed to the original units; Adjusted GMC ratio = 23.2, 95% CI 2-sided [17.9 to 30]

2. Primary Outcome: Anti-Varicella Zoster Virus (VZV) gE Antibody Concentrations
Description: Antibody concentrations as determined by ELISA are presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL). The seropositivity cut-off value was greater than or equal to (≥) 97 mIU//mL.
Time Frame: At Month 2
Population: The analysis was performed on the ATP cohort for Humoral immunogenicity which included all evaluable subjects for which the active phase time point Month 2 data were obtained from the ATP cohort for Humoral Immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 87 | 98
mIU/mL | 18291.7 [14432.1 to 23183.5] | 1060.5 [873.9 to 1287.1]

3. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal every day activities. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of study vaccine administered, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 112 | 110
Participants
  Any Pain, Dose 1 | 83 | 2
  Grade 3 Pain, Dose 1 | 8 | 0
  Any Redness, Dose 1 | 33 | 0
  Grade 3 Redness, Dose 1 | 2 | 0
  Any Swelling, Dose 1 | 15 | 1
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 98 | 105
  Any Pain, Dose 2 | 52 | 5
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 98 | 105
  Grade 3 Pain, Dose 2 | 4 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 98 | 105
  Any Redness, Dose 2 | 20 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 98 | 105
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 98 | 105
  Any Swelling, Dose 2 | 8 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 98 | 105
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Across doses | 90 | 7
  Grade 3 Pain, Across doses | 11 | 0
  Any Redness, Across doses | 40 | 0
  Grade 3 Redness, Across doses | 2 | 0
  Any Swelling, Across doses | 18 | 1
  Grade 3 Swelling, Across doses | 0 | 0

4. Primary Outcome: Number of Days With Solicited Local Symptoms
Description: The number of days with any local symptoms has been assessed during the post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses with the symptom
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 112 | 110
Number analyzed (Doses with the symptom) | 83 | 5
Days
  Pain, Dose 1: number analyzed (Doses with the symptom) | 8 | 2
  Pain, Dose 1 | 2.0 [2.0 to 4.0] | 2.0 [1.0 to 3.0]
  Pain, Dose 2: number analyzed (Participants) | 98 | 105
  Pain, Dose 2: number analyzed (Doses with the symptom) | 52 | 5
  Pain, Dose 2 | 2.0 [1.0 to 3.5] | 1.0 [1.0 to 2.0]
  Redness, Dose 1: number analyzed (Doses with the symptom) | 33 | 0
  Redness, Dose 1 | 3.0 [2.0 to 5.0] |
  Redness, Dose 2: number analyzed (Participants) | 98 | 105
  Redness, Dose 2: number analyzed (Doses with the symptom) | 20 | 0
  Redness, Dose 2 | 4.0 [2.0 to 5.0] |
  Swelling, Dose 1: number analyzed (Doses with the symptom) | 15 | 1
  Swelling, Dose 1 | 4.0 [2.0 to 5.0] | 7.0 [7.0 to 7.0]
  Swelling, Dose 2: number analyzed (Participants) | 98 | 105
  Swelling, Dose 2: number analyzed (Doses with the symptom) | 8 | 0
  Swelling, Dose 2 | 3.5 [2 to 5.5] |

5. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal [symptoms included nausea, vomiting, diarrhoea and/or abdominal pain], headache, myalgia, shivering and fever [defined as oral, axillary or tympanic temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 112 | 110
Participants
  Any Fatigue, Dose 1 | 56 | 44
  Grade 3 Fatigue, Dose 1 | 10 | 3
  Related Fatigue, Dose 1 | 15 | 10
  Any Gastrointestinal, Dose 1 | 32 | 21
  Grade 3 Gastrointestinal, Dose 1 | 2 | 5
  Related Gastrointestinal, Dose 1 | 9 | 2
  Any Headache, Dose 1 | 28 | 24
  Grade 3 Headache, Dose 1 | 3 | 1
  Related Headache, Dose 1 | 10 | 4
  Any Myalgia, Dose 1 | 50 | 17
  Grade 3 Myalgia, Dose 1 | 8 | 3
  Related Myalgia, Dose 1 | 25 | 3
  Any Shivering, Dose 1 | 27 | 13
  Grade 3 Shivering, Dose 1 | 5 | 2
  Related Shivering, Dose 1 | 12 | 4
  Any Fever, Dose 1 | 13 | 4
  Grade 3 Fever, Dose 1 | 0 | 0
  Related Fever, Dose 1 | 11 | 1
  Any Fatigue, Dose 2: number analyzed (Participants) | 97 | 104
  Any Fatigue, Dose 2 | 57 | 57
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 97 | 104
  Grade 3 Fatigue, Dose 2 | 9 | 6
  Related Fatigue, Dose 2: number analyzed (Participants) | 97 | 104
  Related Fatigue, Dose 2 | 6 | 8
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 97 | 104
  Any Gastrointestinal, Dose 2 | 41 | 39
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 97 | 104
  Grade 3 Gastrointestinal, Dose 2 | 5 | 3
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 97 | 104
  Related Gastrointestinal, Dose 2 | 6 | 2
  Any Headache, Dose 2: number analyzed (Participants) | 97 | 104
  Any Headache, Dose 2 | 29 | 25
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 97 | 104
  Grade 3 Headache, Dose 2 | 3 | 2
  Related Headache, Dose 2: number analyzed (Participants) | 97 | 104
  Related Headache, Dose 2 | 7 | 2
  Any Myalgia, Dose 2: number analyzed (Participants) | 97 | 104
  Any Myalgia, Dose 2 | 32 | 23
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 97 | 104
  Grade 3 Myalgia, Dose 2 | 4 | 1
  Related Myalgia, Dose 2: number analyzed (Participants) | 97 | 104
  Related Myalgia, Dose 2 | 13 | 4
  Any Shivering, Dose 2: number analyzed (Participants) | 97 | 104
  Any Shivering, Dose 2 | 20 | 17
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 97 | 104
  Grade 3 Shivering, Dose 2 | 3 | 1
  Related Shivering, Dose 2: number analyzed (Participants) | 97 | 104
  Related Shivering, Dose 2 | 6 | 4
  Any Fever, Dose 2: number analyzed (Participants) | 97 | 104
  Any Fever, Dose 2 | 8 | 1
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 97 | 104
  Grade 3 Fever, Dose 2 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 97 | 104
  Related Fever, Dose 2 | 4 | 0
  Any Fatigue, Across doses | 78 | 68
  Grade 3 Fatigue, Across doses | 16 | 8
  Related Fatigue, Across doses | 19 | 14
  Any Gastrointestinal, Across doses | 51 | 49
  Grade 3 Gastrointestinal, Across doses | 6 | 7
  Related Gastrointestinal, Across doses | 11 | 3
  Any Headache, Across doses | 43 | 40
  Grade 3 Headache, Across doses | 6 | 3
  Related Headache, Across doses | 16 | 6
  Any Myalgia, Across doses | 60 | 31
  Grade 3 Myalgia, Across doses | 12 | 4
  Related Myalgia, Across doses | 30 | 5
  Any Shivering, Across doses | 39 | 25
  Grade 3 Shivering, Across doses | 6 | 3
  Related Shivering, Across doses | 16 | 5
  Any Temperature, Across doses | 20 | 5
  Grade 3 Temperature, Across doses | 0 | 0
  Related Temperature, Across doses | 14 | 1

6. Primary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with any general symptoms has been assessed during the post-vaccination period.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Doses with the symptom
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 112 | 110
Number analyzed (Doses with the symptom) | 57 | 57
Days
  Fatigue, Dose 1: number analyzed (Doses with the symptom) | 56 | 44
  Fatigue, Dose 1 | 3.0 [1.5 to 6.0] | 5.0 [2.0 to 6.0]
  Fatigue, Dose 2: number analyzed (Participants) | 97 | 104
  Fatigue, Dose 2 | 5.0 [2.0 to 7.0] | 5.0 [3.0 to 7.0]
  Gastrointestinal symptoms, Dose 1: number analyzed (Doses with the symptom) | 32 | 21
  Gastrointestinal symptoms, Dose 1 | 2.5 [1.5 to 4.0] | 4.0 [2.0 to 6.0]
  Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 97 | 104
  Gastrointestinal symptoms, Dose 2: number analyzed (Doses with the symptom) | 41 | 39
  Gastrointestinal symptoms, Dose 2 | 4.0 [3.0 to 7.0] | 3.0 [2.0 to 7.0]
  Headache, Dose 1: number analyzed (Doses with the symptom) | 28 | 24
  Headache, Dose 1 | 2.0 [1.0 to 3.5] | 2.0 [1.5 to 4.5]
  Headache, Dose 2: number analyzed (Participants) | 97 | 104
  Headache, Dose 2: number analyzed (Doses with the symptom) | 29 | 25
  Headache, Dose 2 | 2.0 [2.0 to 6.0] | 2.0 [1.0 to 5.0]
  Myalgia, Dose 1: number analyzed (Doses with the symptom) | 50 | 17
  Myalgia, Dose 1 | 2.5 [1.0 to 4.0] | 2.0 [2.0 to 6.0]
  Myalgia, Dose 2: number analyzed (Participants) | 97 | 104
  Myalgia, Dose 2: number analyzed (Doses with the symptom) | 32 | 23
  Myalgia, Dose 2 | 3.0 [2.0 to 5.5] | 5.0 [3.0 to 7.0]
  Shivering, Dose 1: number analyzed (Doses with the symptom) | 27 | 13
  Shivering, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0]
  Shivering, Dose 2: number analyzed (Participants) | 97 | 104
  Shivering, Dose 2: number analyzed (Doses with the symptom) | 20 | 17
  Shivering, Dose 2 | 3.0 [1.0 to 6.0] | 2.0 [1.0 to 4.0]
  Temperature, Dose 1: number analyzed (Doses with the symptom) | 13 | 4
  Temperature, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Temperature, Dose 2: number analyzed (Participants) | 97 | 104
  Temperature, Dose 2: number analyzed (Doses with the symptom) | 8 | 1
  Temperature, Dose 2 | 1.5 [1.0 to 2.5] | 1.0 [1.0 to 1.0]

7. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 117 | 115
Participants
  Any AE(s) | 100 | 103
  Grade 3 AE(s) | 18 | 15
  Related AE(s) | 10 | 9

8. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Related SAE= SAE assessed by the investigator as causally related to the study vaccination.
Time Frame: From first dose up to 30 days post last vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 117 | 115
Participants
  Any SAEs | 16 | 14
  Related SAEs | 0 | 0

9. Primary Outcome: Number of Subjects With Any and Related Potential Immune Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Related = pIMDs assessed by the investigator as causally related to the study vaccination.
Time Frame: From first vaccination up to 30 days post last vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 117 | 115
Participants
  Any pIMDs | 0 | 0
  Related pIMDs | 0 | 0

10. Secondary Outcome: Anti-VZV gE Antibody Concentrations
Description: as for outcome 2
Time Frame: At Months 0, 1, 6 and 13
Population: The analysis was performed on the Adapted ATP cohort for Humoral immunogenicity which included all evaluable subjects for which the active phase time points Months 0, 1 and 2 data were obtained from the ATP cohort for Humoral Immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 87 | 97
mIU/mL
  Anti-VZV gE, Month 0: number analyzed (Participants) | 87 | 94
  Anti-VZV gE, Month 0 | 1049.8 [865.8 to 1273.0] | 1116.7 [918.4 to 1358.0]
  Anti-VZV gE, Month 1: number analyzed (Participants) | 85 | 97
  Anti-VZV gE, Month 1 | 24793.1 [18747.8 to 32787.6] | 1107.2 [920.0 to 1332.6]
  Anti-VZV gE, Month 6: number analyzed (Participants) | 42 | 43
  Anti-VZV gE, Month 6 | 7730.4 [5358.4 to 11152.2] | 1380.2 [1066.3 to 1786.6]
  Anti-VZV gE, Month 13: number analyzed (Participants) | 68 | 70
  Anti-VZV gE, Month 13 | 4477.3 [3482.4 to 5756.3] | 1064.7 [845.9 to 1340.1]

11. Secondary Outcome: Number of Subjects With Vaccine Responses for Anti-gE Antibody ELISA Concentrations
Description: Vaccine response defined as: For initially seronegative subjects, antibody concentration at post-vaccination ≥ 4 fold the cut-off for Anti-gE (4x97 mIU/ml); For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration.
Time Frame: At Months 1, 2, 6 and 13
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 87 | 94
Participants
  Vaccine responders Month 1: number analyzed (Participants) | 85 | 93
  Vaccine responders Month 1 | 73 | 0
  Vaccine responders Month 2 | 75 | 0
  Vaccine responders Month 6: number analyzed (Participants) | 42 | 42
  Vaccine responders Month 6 | 31 | 1
  Vaccine responders Month 13: number analyzed (Participants) | 68 | 69
  Vaccine responders Month 13 | 35 | 0

12. Secondary Outcome: Descriptive Statistics of the Frequency of gE-specific CD4[2+] T-cells in PreChemo Groups
Description: Descriptive statistics were tabulated for CD4[2+] cells, which are gE specific CD4+ T-cells with at least two activation markers ([2+]), expressed from the activation markers interferon-gamma (IFN-γ), interleukin-2 (IL-2), tumour necrosis factor-alpha (TNF-α) and cluster of differentiation 40-ligand (CD40-L), as determined by intracellular cytokine staining (ICS) method.
Time Frame: At Months 0, 1, 2 and 13
Population: The analysis was performed on the PreChemo groups from the Adapted ATP cohort for Cell Mediated Immunity (CMI) immunogenicity which included all evaluable subjects for which the active phase time points Months 0, 1 and 2 data were obtained from the ATP cohort for CMI immunogenicity.
Measure: Median (Inter-Quartile Range); unit: CD4 T-cells/million T-cells
Arm/Group | GSK1437173A-PreChemo | Placeb-PreChemo
Number analyzed (Participants) | 25 | 30
CD4 T-cells/million T-cells
  CD4[2+] T-cells, Month 0: number analyzed (Participants) | 25 | 27
  CD4[2+] T-cells, Month 0 | 127.3 [49.7 to 192.4] | 104.8 [27.5 to 151.5]
  CD4[2+] T-cells, Month 1 | 391.9 [139.7 to 603.7] | 50.0 [1.0 to 179.4]
  CD4[2+] T-cells, Month 2: number analyzed (Participants) | 22 | 29
  CD4[2+] T-cells, Month 2 | 778.8 [393.1 to 1098.2] | 61.8 [17.4 to 139.5]
  CD4[2+] T-cells, Month 13: number analyzed (Participants) | 18 | 19
  CD4[2+] T-cells, Month 13 | 332.9 [114.9 to 604.6] | 51.2 [1.0 to 288.6]

13. Secondary Outcome: Number of Subjects With Vaccine Responses for gE-specific CD4[2+] T-cells in PreChemo Groups
Description: Vaccine response defined as: For initially seronegative subjects with pre-vaccination T-cell frequencies below the threshold, at least a 2-fold increase as compared to the threshold (2x320 Events/10E6 CD4+ T cells); For initially seropositive subjects with pre-vaccination T-cell frequencies above the threshold, at least a 2-fold increase as compared to pre-vaccination T-cell frequencies.
Time Frame: At Months 1, 2 and 13
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A-PreChemo | Placeb-PreChemo
Number analyzed (Participants) | 25 | 27
Participants
  CD4[2+] T-cells, Month 1 | 5 | 0
  CD4[2+] T-cells, Month 2: number analyzed (Participants) | 22 | 27
  CD4[2+] T-cells, Month 2 | 11 | 0
  CD4[2+] T-cells, Month 13: number analyzed (Participants) | 17 | 16
  CD4[2+] T-cells, Month 13 | 3 | 0

14. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Related SAE = SAE assessed by the investigator as causally related to the study vaccination.
Time Frame: From 30 days post last vaccination up to study end (Month 13)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 117 | 115
Participants
  Any SAEs | 30 | 31
  Related SAEs | 0 | 0

15. Secondary Outcome: Number of Subjects With Any Potential Immune Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From 30 days post last vaccination up to study end (Month 13)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 117 | 115
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during the 30-day (Days 0-29) post-vaccination period; SAEs: from first dose up to study end (Month 13).
Arm/Group | GSK1437173A Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 12/117 | 11/115
Serious Adverse Events (participants affected / at risk) | 36/117 | 42/115
Other Adverse Events (participants affected / at risk) | 113/117 | 103/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=117) | Placebo Group (N=115)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (8) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (2) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Hepatitis c (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 2 (3)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Gastrostomy failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=117) | Placebo Group (N=115)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (21) | 23 (23)
Asthenia (General disorders) | 30 (34) | 28 (32)
Chills (General disorders) | 39 (48) | 25 (30)
Constipation (Gastrointestinal disorders) | 16 (19) | 11 (11)
Decreased appetite (Metabolism and nutrition disorders) | 9 (12) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 9 (12) | 10 (10)
Dysgeusia (Nervous system disorders) | 1 (1) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 13 (13)
Erythema (Skin and subcutaneous tissue disorders) | 43 (58) | 1 (1)
Fatigue (General disorders) | 80 (118) | 69 (109)
Gastrointestinal disorder (Gastrointestinal disorders) | 51 (74) | 51 (63)
Headache (Nervous system disorders) | 45 (61) | 41 (52)
Mucosal inflammation (General disorders) | 9 (11) | 6 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 62 (88) | 33 (45)
Nausea (Gastrointestinal disorders) | 31 (36) | 28 (33)
Neutropenia (Blood and lymphatic system disorders) | 11 (12) | 14 (16)
Pain (General disorders) | 90 (139) | 7 (7)
Pyrexia (General disorders) | 22 (23) | 9 (9)
Swelling (General disorders) | 18 (23) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (10) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.